CLINICAL TRIAL: NCT04475016
Title: A Single Center and Single Arm Study of TIP (Paclitaxel + Ifosfamide + Cisplatin) Combined With Nimotuzumab & Triprilimab as Neoadjuvant Treatment in Locally Advanced Penile Cancer
Brief Title: TIP (Paclitaxel + Ifosfamide + Cisplatin) Combined With Nimotuzumab & Triprilimab as Neoadjuvant Treatment in Locally Advanced Penile Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Director, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-103-01
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Penile Cancer
MeSH Terms: conditions — Penile Neoplasms | interventions — Albumin-Bound Paclitaxel; Ifosfamide; Cisplatin; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Therapy (Experimental): TIP (Paclitaxel + Ifosfamide + Cisplatin) & Nimotuzumab & Triprilimab
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Ifosfamide; Drug: Cisplatin; Drug: Nimotuzumab; Drug: Triprilimab

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel — 260 mg/m² IV over 30 minutes on Day 1
Drug: Ifosfamide — 1200 mg/m² IV over 2 hours on Days 1-3
Drug: Cisplatin — 25 mg/m² IV over 2 hours on Days 1-3
Drug: Nimotuzumab — 400 mg IV on Day 1
Drug: Triprilimab — 240 mg IV on Day 1

SUMMARY:
Primary Objective:To evaluate the efficacy and safety of TIP (paclitaxel + ifosfamide + cisplatin) combined with nimotuzumab & triprilimab as neoadjuvant treatment in locally advanced penile cancer.

DETAILED DESCRIPTION:
Penile cancer is a rare malignant tumor, which often occurs in the inner plate of prepuce and glans. Squamous cell carcinoma is the most common pathological type. Lymph node metastasis is a crucial factor that leads to poor prognosis of penile cancer. The 5-year OS of penile cancer patients without lymph node metastasis is 90%. Still, it goes down sharply in patients with inguinal lymph node metastasis and pelvic lymph node metastasis, which is 50% and 0%, respectively.

Using neoadjuvant chemotherapy to treat patients with locally advanced penile cancer (T4, any N stage, or any T stage, N3) may improve their prognosis. TIP (Paclitaxel + Ifosfamide + Cisplatin) regimen is the first line neoadjuvant treatment recommended by NCCN guidelines. Epidermal growth factor receptor (EGFR) plays a vital role in the development of penile cancer. It's also an important therapeutic target for penile cancer. PD-1 is an immune checkpoint molecule on the surface of T cells. In recent years, immune-checkpoint inhibitors targeting PD-1 have shown good efficacy in a variety of tumors. Some phase II / III clinical trials have shown that PD-1 inhibitors can improve the prognosis of patients with lung squamous cell carcinoma, head and neck squamous cell carcinoma and cervical cancer. Previous studies have found that PD-L1 is highly expressed in 40% - 60% of penile cancer, suggesting that penile cancer patients may benefit from immunotherapy.

The management of penile cancer with lymph node metastasis is difficult, especially for N2-3 stage. This phase II study aim to explore an effective combination therapy for locally advanced penile cancer. 29 patients need to be enrolled.TIP & nimotuzumab & triprilimab will be administered per 21-day until surgery, evidence of disease progression or onset of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinoma confirmed by histology or cytology;
2. Clinical Stage is Locally advanced penile cancer (T4, any N stage; or any T stage, N3);
3. No prior chemotherapy for newly diagnosed or relapsed patients;
4. There is at least one measurable lesion according to the solid tumor efficacy evaluation standard RECIST1.1;
5. the Eastern Cooperative Oncology Group (ECOG) scored 0-2;
6. Blood marrow function: Hemoglobin(Hb) >/= 80g/L; White blood cell count >/= 3.0x10^9/L; Neutrophil count >/= 1.5x10^9/L; Platelet count >/= 100x10^9/L;
7. Liver function: AST, ALT, ALP </= 2.5 ULN; Total bilirubin </= 1.5 ULN;
8. Estimated survival >/= 12 months;
9. No prior serious disease history of systemic organ;
10. The participant unterstand this study procedure and sign the informed consent.

Exclusion Criteria:

1. Peripheral neuropathy degree >/=2 (affecting patient's function);
2. Previously received any other experimental drug treatment within 4 weeks before enrollment;
3. Patients with other cancer at present, or have other malignent tumor history within past 5 years. Except for: (1) Cured skin non-malignant melanoma; (2) Curable tumor, including low-risk prostate cancer (T1a, Gleason score<6, PSA<0.5ng/ml), superficial bladder cancer and so on; (3) Other solid tumors have received radical treatment, and no recurrence or metastasis has been found at least 5 years;
4. Other serious or poorly controlled concomitant diseases, including but not limited to: (1) Severe or acute attack disease history of cardiovascular, liver, respiratory, kidney, blood ,endocrine or neuropsychiatric system within 6 months; (2) Active infection history and needed antibiotic treatment within 2 weeks before enrollment; (3) Congestive heart failure (grade III-IV); (4) Unstable angina pectoris or myocardial infarction history within 6 months.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Pathologically Complete Response | 12 weeks
  Histopathologic assessment for patients undergoing surgical resection followed by 4 cycles of neoadjuvant treatment. Pathologically complete response is defined as the absence of noninvasive tumor residuals in inguinal lymph node and pelvic lymph node after neoadjuvant chemotherapy as assessed by American Joint Committee on Cancer (AJCC) staging version 8.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks
  ORR is defined as the percentage of participants who achieved a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression Free Survival (PFS) | 2 months
  Progression free survival is defined as the time from the randomization to tumor progression or death due to any cause.
Overall Survival (OS) | 6 months
  Overall survival is defined as the time from randomization to death due to any cause.
Adverse events | 2-months
  Number of participants with treatment-related adverse events as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China